CLINICAL TRIAL: NCT04651842
Title: Impact of Acute Insulin Resistance on Myocardial Blush in Non- Diabetic Patients Undergoing Primary Percutaneous Coronary Intervention
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Soher Moustafa Kasem, Prof, Assiut University
Other Study IDs: Insulin resistance and PCI
Record Dates: First submitted 2020-11-26; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Insulin Resistance and PCI
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HOMA IR high: classified based on equal tertile of HOMA IR level into 3 equal groups ( high>6.6)
  Interventions: Device: PCI
- HOMA IR intermediate: classified based on equal tertile of HOMA IR level into 3 equal groups ( intermediate 4.6-6.6, )
  Interventions: Device: PCI
- HOMA IR low: classified based on equal tertile of HOMA IR level into 3 equal groups (low ≤ 4.6, )
  Interventions: Device: PCI

INTERVENTIONS:
Device: PCI — Acute Insulin Resistance on Myocardial Blush in Non- Diabetic Patients Undergoing Primary Percutaneous Coronary Intervention
  Other Names: primary Insulin resistance

SUMMARY:
Full myocardial reperfusion with restoration of coronary microcirculatory function (CMF) is a therapeutic goal in ST-segment elevation myocardial infarction (STEMI).1 Despite the success of primary percutaneous coronary intervention (pPCI), it is not achieved in 30% to 50% of patients.2,3 Insulin resistance (IR) as a part of metabolic syndrome is an important risk factor for the development of cardiac and vascular impairments and carries ominous prognosis in the setting of acute myocardial infarction.4 As a part of metabolic syndrome, IR is associated with myocardial and microvascular injury after STEMI in clinical studies. As phenomenon per se, independent of other components of metabolic syndrome, IR was related to ischemic myocardial injury after elective PCI.5

Recently, IR in the early phase of acute coronary syndrome in non-diabetic patients, assessed by the homeostatic model assessment (HOMA) index, was established as an independent predictor of in-hospital mortality. This "acute" IR is a part of the acute glycometabolic response to stress, can be transient and can occur even in patients without chronic glycometabolic derangements.6

Acute IR comprises acute hyperglycemia and/or acute hyperinsulinemia; Hyperglycemia has the prognostic relevance of hyperinsulinemia in STEMI patients and its relationship with coronary flow are less well evaluated.it also acknowledged direct acute negative cardiovascular effects as it is contributing to incomplete myocardial reperfusion and CMF impairment. The prognostic relevance of hyperinsulinemia in STEMI patients and its relationship with coronary flow are less well evaluated and acknowledged.7,8 Myocardial blush was first defined by Arnoud van't Hof etal . It is a qualitative visual assessment of the amount of contrast medium filling a territory supplied by a pericardial coronary artery.9 Myocardial blush grade is a valuable tool for assessing coronary microvasculature and myocardial perfusion in patients undergoing coronary angiography and angioplasty.

Reduced myocardial blush grade identifies patients at higher risk who need more aggressive treatment both during the procedure to improve myocardial perfusion and later for secondary prevention.10

We postulate that IR can occur in the early post pPCI period as a dynamic phenomenon even in non-diabetic patients, and be related to the development of microvascular injury. We have defined myocardial blush as a marker of coronary microvascular function, Accordingly, we have evaluated IR in relation to myocardial blush in non-diabetic STEMI patients treated by pPCI. as a primary end-point. The residual ST-segment elevation, post-TFC%; and MACE were secondary end points. The HOMA index is a simple and inexpensive marker of IR primary used in chronic states. It was recently validated against euglycemic hyperinsulinemic clamp in STEMI patients as feasible for assessing IR during myocardial infarction and therefore used in the current study.11

DETAILED DESCRIPTION:
Myocardial blush grade is valuable tool for assessing coronary microvasculature and myocardial perfusion in patients undergoing coronary angiography and angioplasty and its reduction identifies patients at high risk. In this study we investigate the association of acute insulin resistance with myocardial blush grade and outcome in non-diabetic patients with ST-segment elevation myocardial infarction (STEMI).

ELIGIBILITY:
Inclusion Criteria:

* This cross-sectional comparative study included 240 non-diabetic patients with acute STEMI of both sexes and different ages selected from cardiology department in Assiut University Hospital who underwent primary percutaneous coronary intervention (PCI) between first of May 2018 and first of May 2019.

Exclusion Criteria:

* Patients were excluded from this study if they had diabetes mellitus; renal insufficiency (creatinine >2 mg/dl); advanced hepatic dysfunction; taken anti-oxidant supplement/therapy within the past 4 weeks before enrollment; pregnant; were alcoholic; had allergy to radiographic contrast; uncooperative patient or patient refusal; also if they had malignancy; chronic heart failure or cardiomyopathy; prior myocardial infarction and diseases requiring steroid therapy

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 240 non-diabetic patients with acute STEMI of both sexes and different ages selected from cardiology department in Assiut University Hospital who underwent primary percutaneous coronary intervention (PCI) between first of May 2018 and first of May 2019.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
arrythmia,LVF,Pulmonary edema,Cardiogenic shock, In hospital re-infarction,In hospital stent thrombosis | May2018 to May 2019

SECONDARY OUTCOMES:
In hospial mortality | May 2018 to May2019

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Asyut, Egypt

REFERENCES:
- [Background] Lerman A, Holmes DR, Herrmann J, Gersh BJ. Microcirculatory dysfunction in ST-elevation myocardial infarction: cause, consequence, or both? Eur Heart J. 2007 Apr;28(7):788-97. doi: 10.1093/eurheartj/ehl501. Epub 2007 Mar 8. PMID 17347176
- [Background] Niccoli G, Burzotta F, Galiuto L, Crea F. Myocardial no-reflow in humans. J Am Coll Cardiol. 2009 Jul 21;54(4):281-92. doi: 10.1016/j.jacc.2009.03.054. PMID 19608025
- [Background] Arnold SV, Lipska KJ, Li Y, Goyal A, Maddox TM, McGuire DK, Spertus JA, Kosiborod M. The reliability and prognosis of in-hospital diagnosis of metabolic syndrome in the setting of acute myocardial infarction. J Am Coll Cardiol. 2013 Aug 20;62(8):704-8. doi: 10.1016/j.jacc.2013.02.062. Epub 2013 Apr 3. PMID 23563136
- [Background] Uetani T, Amano T, Harada K, Kitagawa K, Kunimura A, Shimbo Y, Harada K, Yoshida T, Kato B, Kato M, Marui N, Nanki M, Hotta N, Ishii H, Matsubara T, Murohara T. Impact of insulin resistance on post-procedural myocardial injury and clinical outcomes in patients who underwent elective coronary interventions with drug-eluting stents. JACC Cardiovasc Interv. 2012 Nov;5(11):1159-67. doi: 10.1016/j.jcin.2012.07.008. PMID 23174640
- [Background] Sanjuan R, Blasco ML, Huerta R, Palacios L, Carratala A, Nunyez J, Sanchis J. Insulin resistance and short-term mortality in patients with acute myocardial infarction. Int J Cardiol. 2014 Mar 15;172(2):e269-70. doi: 10.1016/j.ijcard.2013.12.207. Epub 2014 Jan 8. No abstract available. PMID 24485226
- [Background] Zarich SW, Nesto RW. Implications and treatment of acute hyperglycemia in the setting of acute myocardial infarction. Circulation. 2007 May 8;115(18):e436-9. doi: 10.1161/CIRCULATIONAHA.105.535732. No abstract available. PMID 17485582
- [Background] van 't Hof AW, Liem A, Suryapranata H, Hoorntje JC, de Boer MJ, Zijlstra F. Angiographic assessment of myocardial reperfusion in patients treated with primary angioplasty for acute myocardial infarction: myocardial blush grade. Zwolle Myocardial Infarction Study Group. Circulation. 1998 Jun 16;97(23):2302-6. doi: 10.1161/01.cir.97.23.2302. PMID 9639373
- [Background] Tsvetkov H, Mosseri M. Myocardial blush grade: an interventional method for assessing myocardial perfusion. Isr Med Assoc J. 2008 Jun;10(6):465-7. No abstract available. PMID 18669149
- [Background] Moura FA, Carvalho LS, Cintra RM, Martins NV, Figueiredo VN, Quinaglia e Silva JC, Almeida OL, Coelho OR, Sposito AC. Validation of surrogate indexes of insulin sensitivity in acute phase of myocardial infarction based on euglycemic-hyperinsulinemic clamp. Am J Physiol Endocrinol Metab. 2014 Feb 15;306(4):E399-403. doi: 10.1152/ajpendo.00566.2013. Epub 2013 Dec 17. PMID 24347056
- [Background] American Diabetes Association. Standards of medical care in diabetes--2012. Diabetes Care. 2012 Jan;35 Suppl 1(Suppl 1):S11-63. doi: 10.2337/dc12-s011. No abstract available. PMID 22187469
- [Background] James PA, Oparil S, Carter BL, Cushman WC, Dennison-Himmelfarb C, Handler J, Lackland DT, LeFevre ML, MacKenzie TD, Ogedegbe O, Smith SC Jr, Svetkey LP, Taler SJ, Townsend RR, Wright JT Jr, Narva AS, Ortiz E. 2014 evidence-based guideline for the management of high blood pressure in adults: report from the panel members appointed to the Eighth Joint National Committee (JNC 8). JAMA. 2014 Feb 5;311(5):507-20. doi: 10.1001/jama.2013.284427. PMID 24352797
- [Background] Grundy SM, Cleeman JI, Merz CN, Brewer HB Jr, Clark LT, Hunninghake DB, Pasternak RC, Smith SC Jr, Stone NJ; Coordinating Committee of the National Cholesterol Education Program. Implications of recent clinical trials for the National Cholesterol Education Program Adult Treatment Panel III Guidelines. J Am Coll Cardiol. 2004 Aug 4;44(3):720-32. doi: 10.1016/j.jacc.2004.07.001. PMID 15358046
- [Background] de Boer MJ, Reiber JH, Suryapranata H, van den Brand MJ, Hoorntje JC, Zijlstra F. Angiographic findings and catheterization laboratory events in patients with primary coronary angioplasty or streptokinase therapy for acute myocardial infarction. Eur Heart J. 1995 Oct;16(10):1347-55. doi: 10.1093/oxfordjournals.eurheartj.a060741. PMID 8746902
- [Background] TIMI Study Group. The Thrombolysis in Myocardial Infarction (TIMI) trial. Phase I findings. N Engl J Med. 1985 Apr 4;312(14):932-6. doi: 10.1056/NEJM198504043121437. No abstract available. PMID 4038784
- [Background] Gibson CM, Cannon CP, Daley WL, Dodge JT Jr, Alexander B Jr, Marble SJ, McCabe CH, Raymond L, Fortin T, Poole WK, Braunwald E. TIMI frame count: a quantitative method of assessing coronary artery flow. Circulation. 1996 Mar 1;93(5):879-88. doi: 10.1161/01.cir.93.5.879. PMID 8598078
- [Background] Gibson CM, Cannon CP, Murphy SA, Ryan KA, Mesley R, Marble SJ, McCabe CH, Van De Werf F, Braunwald E. Relationship of TIMI myocardial perfusion grade to mortality after administration of thrombolytic drugs. Circulation. 2000 Jan 18;101(2):125-30. doi: 10.1161/01.cir.101.2.125. PMID 10637197
- [Background] van 't Hof AW, Liem A, de Boer MJ, Zijlstra F. Clinical value of 12-lead electrocardiogram after successful reperfusion therapy for acute myocardial infarction. Zwolle Myocardial infarction Study Group. Lancet. 1997 Aug 30;350(9078):615-9. doi: 10.1016/s0140-6736(96)07120-6. PMID 9288043
- [Background] Nishio K, Shigemitsu M, Kusuyama T, Fukui T, Kawamura K, Itoh S, Konno N, Katagiri T. Insulin resistance in nondiabetic patients with acute myocardial infarction. Cardiovasc Revasc Med. 2006 Apr-Jun;7(2):54-60. doi: 10.1016/j.carrev.2005.12.004. PMID 16757401
- [Background] Li L, Messina JL. Acute insulin resistance following injury. Trends Endocrinol Metab. 2009 Nov;20(9):429-35. doi: 10.1016/j.tem.2009.06.004. Epub 2009 Oct 1. PMID 19800814
- [Background] Pretty CG, Le Compte AJ, Chase JG, Shaw GM, Preiser JC, Penning S, Desaive T. Variability of insulin sensitivity during the first 4 days of critical illness: implications for tight glycemic control. Ann Intensive Care. 2012 Jun 15;2(1):17. doi: 10.1186/2110-5820-2-17. PMID 22703645
- [Background] Hedblad B, Nilsson P, Engstrom G, Berglund G, Janzon L. Insulin resistance in non-diabetic subjects is associated with increased incidence of myocardial infarction and death. Diabet Med. 2002 Jun;19(6):470-5. doi: 10.1046/j.1464-5491.2002.00719.x. PMID 12060058
- [Background] Shah RV, Abbasi SA, Heydari B, Rickers C, Jacobs DR Jr, Wang L, Kwong RY, Bluemke DA, Lima JA, Jerosch-Herold M. Insulin resistance, subclinical left ventricular remodeling, and the obesity paradox: MESA (Multi-Ethnic Study of Atherosclerosis). J Am Coll Cardiol. 2013 Apr 23;61(16):1698-706. doi: 10.1016/j.jacc.2013.01.053. PMID 23500236
- [Background] Gruzdeva O, Uchasova E, Dyleva Y, Belik E, Shurygina E, Barbarash O. Insulin resistance and inflammation markers in myocardial infarction. J Inflamm Res. 2013 Jun 17;6:83-90. doi: 10.2147/JIR.S43081. Print 2013. PMID 23837002
- [Background] Lazzeri C, Valente S, Chiostri M, Picariello C, Gensini GF. Correlates of acute insulin resistance in the early phase of non-diabetic ST-elevation myocardial infarction. Diab Vasc Dis Res. 2011 Jan;8(1):35-42. doi: 10.1177/1479164110396744. PMID 21262869
- [Background] Lazzeri C, Sori A, Chiostri M, Gensini GF, Valente S. Prognostic role of insulin resistance as assessed by homeostatic model assessment index in the acute phase of myocardial infarction in nondiabetic patients submitted to percutaneous coronary intervention. Eur J Anaesthesiol. 2009 Oct;26(10):856-62. doi: 10.1097/EJA.0b013e32832a235c. PMID 19367169
- [Background] Timmer JR, Ottervanger JP, de Boer MJ, Dambrink JH, Hoorntje JC, Gosselink AT, Suryapranata H, Zijlstra F, van 't Hof AW; Zwolle Myocardial Infarction Study Group. Hyperglycemia is an important predictor of impaired coronary flow before reperfusion therapy in ST-segment elevation myocardial infarction. J Am Coll Cardiol. 2005 Apr 5;45(7):999-1002. doi: 10.1016/j.jacc.2004.12.050. PMID 15808754
- [Background] L'Huillier I, Zeller M, Mock L, Beer JC, Laurent Y, Sicard P, Vincent-Martin M, Lorgis L, Makki H, Wolf JE, Freysz M, Cottin Y. Relation of hyperglycemia to ST-segment resolution after reperfusion for acute myocardial infarction (from Observatoire des Infarctus de Cote-d'Or Survey [RICO]). Am J Cardiol. 2006 Jul 15;98(2):167-71. doi: 10.1016/j.amjcard.2006.01.087. Epub 2006 May 19. PMID 16828586
- [Derived] Kasem SM, Saied GM, Hegazy ANM, Abdelsabour M. Impact of Acute Insulin Resistance on Myocardial Blush in Non-Diabetic Patients Undergoing Primary Percutaneous Coronary Intervention. Front Cardiovasc Med. 2021 May 10;8:647366. doi: 10.3389/fcvm.2021.647366. eCollection 2021. PMID 34041280